CLINICAL TRIAL: NCT07343570
Title: Comparing Ultrasound-guided Lateral Quadratus Lumborum Block Versus Combined Ilio-inguinal/Ilio-hypogastric /Genitofemoral Block for Postoperative Analgesia After Open Inguinal Hernia Repair: A Double-blind Randomized Controlled Trial
Brief Title: Comparison of Quadratus Lumborum and Combined Groin Nerve Blocks for Postoperative Analgesia After Open Inguinal Hernia Repair.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC. 12.9.2025
Record Dates: First submitted 2025-12-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Analgesia of Inguinal Hernia Repair in Adults
Keywords: Quadratus lumborum [QL] block; Ilioinguinal-iliohypogastric (IIIH) nerve block; Genitofemoral block
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Quadratus lumborum block) (Active Comparator): Ultrasound-guided lateral quadratus lumborum block. Local anesthetic: 30 ml of (Ropivacaine 0.2%) is injected at the appropriate fascial level.
  Interventions: Procedure: Ultrasound-guided lateral quadratus lumborum block
- Group 2 ( Ilio-inguinal and ilio-hypogastric block) (Active Comparator): Ultrasound-guided ilio-inguinal and ilio-hypogastric block. Local anesthesia: 20 ml of 0.2% ropivacaine for ilio-inguinal and ilio-hypogastric block + 10 ml of 0.2% ropivacaine for genitofemoral anaesthesia, total injection volume = 30 ml.
  Interventions: Procedure: Combined ilio-inguinal/ilio-hypogastric/genitofemoral (II-IH-GFN) block

INTERVENTIONS:
Procedure: Ultrasound-guided lateral quadratus lumborum block — Ultrasound-guided lateral quadratus lumborum block. Local anesthetic: 30 ml of (Ropivacaine 0.2%) is injected at the appropriate fascial level.
  Arms: Group 1 (Quadratus lumborum block)
Procedure: Combined ilio-inguinal/ilio-hypogastric/genitofemoral (II-IH-GFN) block — Ultrasound-guided ilio-inguinal and ilio-hypogastric block. Local anesthesia: 20 ml of 0.2% ropivacaine for ilio-inguinal and ilio-hypogastric block + 10 ml of 0.2% ropivacaine for genitofemoral anaesthesia, total injection volume = 30 ml.
  Arms: Group 2 ( Ilio-inguinal and ilio-hypogastric block)

SUMMARY:
This double-blind randomized controlled trial aimes to compares two ultrasound-guided regional techniques-lateral quadratus lumborum block versus combined ilio-inguinal/ilio-hypogastric/genitofemoral (II-IH-GFN) block-for postoperative analgesia after elective unilateral open inguinal hernia repair under spinal anesthesia in adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years.
* ASA physical status I-III.
* Scheduled for elective unilateral open inguinal hernia repair under standardized spinal anesthesia.
* Able to understand and use the Visual Analogue Scale (VAS).
* Provided written informed consent.

Exclusion Criteria:

* Allergy to local anesthetics.
* Coagulopathy or current use of anticoagulants contraindicating peripheral nerve blocks.
* Infection at the injection site.
* Chronic opioid use (daily opioids >2 weeks) or chronic pain syndromes.
* Body mass index (BMI) >40 kg/m².
* Conversion to other surgery or bilateral repair.
* Pregnant patients.
* Refusal to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption in the first 24 hours postoperatively | 24 hours after surgery.
  Measures the total amount of opioid analgesics (expressed as morphine milligram equivalents, MME) consumed during the first postoperative 24 hours. It reflects overall analgesic efficacy of the two block techniques.

SECONDARY OUTCOMES:
Pain intensity (VAS pain scores at rest ) | 24 hours postoperatively.
  Assesses the level of postoperative pain at rest using the Visual Analogue Scale (VAS), where 0 = no pain and 10 = worst imaginable pain.
Pain intensity (VAS pain scores at movement) | 24 hours postoperatively.
  Assesses the level of postoperative pain during movement using the Visual Analogue Scale (VAS), where 0 = no pain and 10 = worst imaginable pain.
Time to first analgesic request | 24 hours.
  Determines the duration of effective analgesia provided by each block, defined as the interval from completion of the block to the first patient request for additional analgesia.
Proportion of patients requiring rescue opioid analgesia | 24 hours.
  Percentage of patients who required additional opioid analgesics beyond the planned postoperative regimen, indicating inadequate analgesia from the primary block.
Incidence of postoperative block-related complications | 24 hours.
  Evaluates safety of the blocks by recording complications such as hematoma, local anesthetic toxicity, or impaired mobility.
Patient satisfaction score | Assessed at 24 hours postoperatively.
  Patient satisfaction with postoperative pain control will be evaluated using a 5-point Likert scale, allowing a simple yet reliable measure of the patient's overall analgesic experience. Each participant will rate their satisfaction as follows: 1 for "very dissatisfied," indicating poor pain relief and marked discomfort; 2 for "dissatisfied," reflecting inadequate but tolerable pain control; 3 for "neutral," representing acceptable analgesia without a clear sense of satisfaction; 4 for "satisfied," denoting good pain relief and minimal discomfort; and 5 for "very satisfied," corresponding to excellent pain control and full contentment with the postoperative analgesia regimen.
Post-anesthesia care unit (PACU) stay duration | 24 hours
  Measures the time spent in the PACU
Total hospital stay duration | 24 hours
  Measures total length of hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared upon a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP